CLINICAL TRIAL: NCT05268068
Title: A Phase 1 Study in Healthy Chinese Subjects to Assess the Pharmacokinetics, Safety and Tolerability After a Single Dose of Risankizumab
Brief Title: A Study of Intravenously (IV) Infused or Subcutaneously (SC) Injected Risankizumab in Healthy Adult Participants in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M17-381
Record Dates: First submitted 2022-03-03; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Risankizumab; ABBV-066; SKYRIZI
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose A of Risankizumab for Subcutaneous (SC) Injection (Experimental): Participants will receive SC injections of risankizumab at dose A and then followed for 140 days.
  Interventions: Drug: Risankizumab
- Dose B of Risankizumab for Subcutaneous (SC) Injection (Experimental): Participants will receive SC injections of risankizumab at dose B and then followed for 140 days.
  Interventions: Drug: Risankizumab
- Dose C of Risankizumab for Intravenous (IV) Infusion (Experimental): Participants will receive IV infusion of risankizumab at dose C and then followed for 140 days.
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Intravenous (IV) Infusion
  Other Names: ABBV-066; SKYRIZI
  Arms: Dose C of Risankizumab for Intravenous (IV) Infusion
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; SKYRIZI
  Arms: Dose A of Risankizumab for Subcutaneous (SC) Injection; Dose B of Risankizumab for Subcutaneous (SC) Injection

SUMMARY:
The objective of this study to assess the pharmacokinetics, safety, tolerability and immunogenicity following a single subcutaneous (SC) or intravenous (IV) dose of risankizumab in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

- Body Mass Index (BMI) is >= 19.0 to <= 26.0 kg/m2 after rounding to the nearest tenth. BMI is calculated as weight in kg divided by the square of height measured in meters.

Exclusion Criteria:

- Previous exposure to any anti-IL-12/23 or anti-IL-23 treatment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-04-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 140 Days
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Maximum Observed Concentration (Cmax) | Up to Approximately 140 Days
  Maximum observed concentration.
Time to Cmax (Tmax) | Up to Approximately 140 Days
  Time to Cmax.
Terminal Phase Elimination Rate Constant (β) | Up to Approximately 140 Days
  Terminal phase elimination rate constant.
Terminal Phase Elimination Half-life (t1/2) | Up to Approximately 140 Days
  Terminal phase elimination half-life.
Area Under the Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) | Up to Approximately 140 Days
  AUC from time 0 to time of the last measurable concentration (AUCt).
AUC from Time 0 to Infinity (AUCinf) | Up to Approximately 140 Days
  AUC from time 0 to infinity (AUCinf).
Apparent Clearance (CL/F) for Subcutaneous (SC) dosing | Up to Approximately 140 Days
  CL/F for SC dosing.
Clearance (CL) for Intravenous (IV) Dosing | Up to Approximately 140 Days
  CL for IV dosing.
Number of Anti-drug antibody (ADA) Titers | Up to Approximately 140 Days
  ADA titers will be tabulated for each participant at the respective study visits.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Shanghai Xuhui Central Hospital /ID# 212830, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No